CLINICAL TRIAL: NCT00952848
Title: The Efficacy of MC5-A ("Scrambler") Therapy in the Management of Chemotherapy-Induced Peripheral Neuropathy: A Phase II Pilot Trial
Brief Title: Electrical Stimulation Therapy Using the MC5-A Scrambler in Reducing Peripheral Neuropathy Caused by Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000644516; MCV-MCC-12110 (Other: VCU Massey Cancer Center)
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Chemotherapeutic Agent Toxicity; Neurotoxicity; Pain; Peripheral Neuropathy; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: pain; neurotoxicity; chemotherapeutic agent toxicity; unspecified adult solid tumor, protocol specific; peripheral neuropathy
MeSH Terms: conditions — Neurotoxicity Syndromes; Pain; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MC5-A Scramble instrument (Experimental): Treatment of chronic neuropathic pain with the MC5-A device
  Interventions: Other: questionnaire administration; Other: Sensory Neuropathy Scale instrument; Other: Quality of Life instrument; Device: MC5-A Scrambler device

INTERVENTIONS:
Other: questionnaire administration — Pain Rating Score
Other: Sensory Neuropathy Scale instrument — ECOG Common Toxicity Criteria for Sensory Neuropathy scale
Other: Quality of Life instrument — Uniscale 0-100 scale global quality of life
Device: MC5-A Scrambler device — Electrical stimulation for 60 minutes

SUMMARY:
RATIONALE: Electronic stimulation using a MC5-A Scrambler may help relieve pain in patients who develop peripheral neuropathy while undergoing chemotherapy treatments for cancer.

PURPOSE: This phase II trial is studying how well MC5-A Scrambler therapy works in reducing peripheral neuropathy caused by chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if MC5-A Scrambler therapy will improve the pain associated with chemotherapy-induced peripheral neuropathy in cancer patients by 20%.

Secondary

* To evaluate the effect of MC5-A therapy on specific pain and neuropathy scales.
* To evaluate the effect of MC5-A therapy on overall quality of life.
* To evaluate the effect of MC5-A therapy on other pain drugs used.
* To evaluate the toxicities of MC5-A therapy.

OUTLINE: Patients undergo gel electrode application on the skin in the most pain-free of the pain-affected area. Patients undergo treatment with the MC5-A Scrambler machine over 60 minutes once daily on days 1-10. On day 1, the treatment intensity is increased every 10 minutes to the maximum intensity individually bearable by the patient without any input of pain or discomfort. The patient should feel the disappearance of the pain during treatment as a sign that the proper nerve pathway(s) has (have) been correctly identified. Subsequent treatments begin at the highest intensity tolerated at the previous treatment. Patients with no improvement after 3 treatments discontinue treatment.

Patients complete questionnaires about symptoms, pain, and quality of life periodically.

After completion of study treatment, patients are followed up at 2 and 4 weeks, monthly for 3 months, and at 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Chemotherapy-induced peripheral neuropathy (CIPN) meeting the following criteria:

  * More than 4 weeks since prior neurotoxic chemotherapy including taxanes (e.g., paclitaxel or docetaxel), platinum-based compounds (e.g., carboplatin, cis-platinum, oxaliplatin), vinca-alkaloids (e.g., vincristine, vinblastine, or vinorelbine), or proteosome inhibitors (e.g., bortezomib)
  * Pain or symptoms of peripheral neuropathy for ≥ 1 month attributed to CIPN
  * Pain stable for ≥ 2 weeks
  * Average daily pain rating of ≥ 5 out of 10 using the pain numerical rating scale (0 is no pain and 10 is worst pain possible)
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of an allergic reaction or intolerance to transcutaneous electronic nerve stimulation
* No pacemaker or implantable drug-delivery system (e.g., Medtronic Synchromed)
* No heart stent or vena cava clips
* No history of epilepsy or brain damage
* No other identified causes of painful paresthesias existing before chemotherapy (e.g., radiation or malignant plexopathy, lumbar or cervical radiculopathy, pre-existing peripheral neuropathy of another etiology [e.g., B12 deficiency, AIDS, monoclonal gammopathy, diabetes, heavy metal poisoning amyloidosis, syphilis, hyperthyroidism, hypothyroidism, inherited neuropathy, etc.])
* No skin conditions (e.g., open sores) that would prevent proper application of the electrodes
* No other medical or other conditions that, in the opinion of the investigators, might compromise the objectives of the study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 30 days since prior and no concurrent investigational agents for pain control
* More than 4 weeks since prior and no concurrent celiac plexus block or other neurolytic pain control treatment
* No prior or concurrent anti-convulsants
* No concurrent neurotoxic or potentially neurotoxic chemotherapy
* Concurrent pain treatments allowed provided the following criteria are met:

  * Pain is not satisfactorily controlled
  * Dose of the other medication has been stable for ≥ 4 weeks

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-06-12; Primary Completion 2009-10 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Smith, MD, Principal Investigator — Massey Cancer Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: 06/12/2009 - 10/26/2009 Location of recruitment: medical clinic
Groups:
- MC5-A Scrambler Instrument: Treatment of chronic neuropathic pain with the MC5-A device
Period: Overall Study
Arm/Group | MC5-A Scrambler Instrument
Started | 18
Completed | 14
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | MC5-A Scrambler Instrument
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score
Description: Change in Neumeric Rating Score for Pain as measured by a Numeric Pain Rating scale between day 0 to day 15.
  Scale is 0 (none) to 10 (severe)
Time Frame: 15 days
Population: Patients treated with MC5A devise for 10 consectuvive days
Measure: Median (90% Confidence Interval); unit: units on a scale
Groups:
- MC5-A Pain Treatment Device: Patients treated with the MC5-A device for chronic chemotherapy-induced peripheral neuropathy
Arm/Group | MC5-A Pain Treatment Device
Number analyzed (Participants) | 14
units on a scale | 2.4 [-3 to 6]

2. Secondary Outcome: Effect of MC5-A on Pain and Neuropathy
Description: Change on pain and neuropathy as measured by the Eastern Cooperative Oncology Group (ECOG) Common Toxicity Criteria for Sensory Neuropathy scale,0=none to 4=paralysis; the World Health Organization (WHO) Classification Scale, 0=none to 4=paralysis; and the Brief Pain Inventory-Short Form, 0=none to 4=most intense pain imaginable. Scores will be averaged.
Time Frame: 2 weeks
Population: Patients treated with MC5A devise for 10 consectuvive days
Measure: Median (90% Confidence Interval); unit: units on a scale
Arm/Group | MC5-A Pain Treatment Device
Number analyzed (Participants) | 14
units on a scale | 1.3 [0.083 to 2.35]

3. Secondary Outcome: Effect of MC5-A on Morphine Oral Equivalent Doses Used Before and After MC5-A Therapy
Description: The change in overal equivalent doses (all narcotic doses will be converted to morphine oral equivalent doses ie as mg/24hours. (All opiates taken will be recorded for the full 24 hours preceding the visit or phone call. All opiates will be converted to the pnmorphine equivalent using the Morphine oral dose equivalents (MOED). The total MOEDs taken during the 24 hours will be the sum of all opiates taken) used before intervention
Time Frame: 2 weeks
Population: Patients treated with MC5A devise for 10 consectuvive days
Measure: Median (90% Confidence Interval); unit: mg/24hr
Arm/Group | MC5-A Pain Treatment Device
Number analyzed (Participants) | 14
mg/24hr | -41.25 [-45.38 to -37.12]

4. Secondary Outcome: Toxicity of MC5-A Therapy on Global Quality of Life Using the Uniscale Instrument
Description: Change on global quality of life. The global quality of life will improve as measured by the Uniscale Linear Analog Scale Assessment (LASA) quality of life scale 0=as bad as it can be to 10=as good as it can be. Scores will be averaged.
Time Frame: 2 weeks
Population: Patients treated with MC5A devise for 10 consectuvive days
Measure: Median (90% Confidence Interval); unit: units on a scale
Arm/Group | MC5-A Pain Treatment Device
Number analyzed (Participants) | 14
units on a scale | 0.08 [0 to 10]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | MC5-A Scrambler Instrument
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MC5-A Scrambler Instrument (N=18)
Seizure (Nervous system disorders) | 1 (1) — Unrelated to intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes